CLINICAL TRIAL: NCT03050645
Title: Diabetes, Metabolic Risk Factors, Autoimmunity and Self-reported Life Style Factors in Women With Previous Gestational Diabetes Mellitus (GDM)
Brief Title: Metabolic Risk and Life Style Factors in Women With Previous Gestational Diabetes Mellitus (GDM)
Status: Completed | Type: Observational
Sponsor: University of Southern Denmark (Other)
Responsible Party: Sponsor
Other Study IDs: University of Southern Denmark
Record Dates: First submitted 2017-01-04; First posted 2017-02-13 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2017-11

CONDITIONS: Type2 Diabetes; Gestational Diabetes; Life Style
MeSH Terms: conditions — Diabetes, Gestational

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood samples
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- previous GDM: Women with previous GDM
- no previous GDM: Women without previous GDM matched on age, pregestational body mass index end time of pregnancy.

SUMMARY:
Women with previous Gestational Diabetes Mellitus (GDM) are characterized by several metabolic abnormalities i.e. insulin resistance, beta-cell dysfunction and increased risk of later Diabetes Mellitus (DM). These latent disorders of glucose metabolism are demasked by the metabolic stress of pregnancy and as a routine, clinical assessment and measurement of HbA1c in addition to an oral glucose tolerance test (OGTT) is offered 3 months post partum.

In this study, women with previous GDM and a control group matched on age, time of birth and BMI around 8 years after pregnancy will be investigated. Information from pregnancy and post partum examination (GDM only) will be used to identify risk factors for later development of DM. Further, life-style factors and mental health according to diabetes status will be studied.

DETAILED DESCRIPTION:
Background

It is well established that women with previous GDM are characterized by several metabolic abnormalities i.e. insulin resistance, beta-cell dysfunction and increased risk of later Diabetes Mellitus (DM). Furthermore, GDM is a heterogeneous condition covering both women with a strong genetic disposition to type 2 DM, women in the early stages of autoimmune DM and rare cases of monogenetic DM. These latent disorders of glucose metabolism are damasked by the metabolic stress of pregnancy.

Aims

1. To study predictors of DM and pre-DM after GDM: a) At the time of pregnancy: age, blood pressure, pre-pregnancy Body Mass Index (BMI), b) 3 months post partum: indices of insulin sensitivity and beta-cell function, lipid profile, GAD-autoantibodies, HbA1c
2. To study lifestyle factors 7-8 years after GDM pregnancy in relation to current diabetes status

Materials and methods

During 2011-2017 women with previous GDM and a control group are invited to a long-term follow-up. Data collection is performed 7-8 years after pregnancy. GDM subjects (n~150), controls (n~50):

1. Anthropometrics: weight, height, waist circumference, blood pressure and length
2. Analyses: p-glucose, s-insulin at 0, 30 and 120 minutes during a 2-h 75 g OGTT. Fasting: total cholesterol, HDL, LDL triglycerides, GAD- autoantibodies, Hba1C, Urine albumin/creatinine ratio.
3. Questionnaires: Information on lifestyle and health status

Data available around pregnancy

Pregnancy data from hospital journals (GDM subjects and controls):

Examinations 3 months post-partum (GDM subjects only):

Clinical examination, 2-h 75 g OGTT with measurements of p-glucose and s- insulin at 0, 30 and 120 minutes, fasting total cholesterol, HDL, LDL and triglycerides, HbA1c and GAD- autoantibodies.

Perspectives

Our current population is unique as clinical, metabolic and autoimmune markers were determined prospectively a few months after GDM pregnancy and at follow-up. Hopefully, the results will enable us to target preventive actions in women with previous GDM and improve our understanding of pathophysiologic mechanisms in pre-diabetic conditions.

ELIGIBILITY:
Inclusion Criteria:

* Previous GDM with information from post partum OGTT
* Danish speaking

Exclusion Criteria:

* Bariatric surgery
* Poorly controlled psychiatric disorder

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: 1. Women with gestational diabetes in a previous pregnancy and information from post partum ogtt.
  2. A control Group of women without GDM matched on pre-pregnancy BMI, age and time of birth.
Sampling Method: Non-Probability Sample
Enrollment: 210 (Actual)
Dates: Start 2011-06; Primary Completion 2017-08 (Actual); Study Completion 2017-08 (Actual)

PRIMARY OUTCOMES:
Type 2 diabetes | 7 to 8 years after giving birth

SECONDARY OUTCOMES:
Plasma glucose (mmol/l) at 0, 30 and 120 minutes during oral glucose tolerance test | 7 to 8 years after giving birth
Serum insulin (mU/l) at 0, 30 and 120 minutes during oral glucose tolerance test | 7 to 8 years after giving birth
Body mass index (kg/m2) | 7 to 8 years after giving birth
Blood pressure (mmHg) | 7 to 8 years after giving birth
Questionnaires, quality of life (SF12), physical and mental summary scores | 7 to 8 years after giving birth
Questionnaires, mental health (WHO-5), WHO-Five well being index | 7 to 8 years after giving birth
Questionnaires, physical activity (PAS 2), physical activity score | 7 to 8 years after giving birth

CONTACTS AND LOCATIONS:
Overall Officials: Dorte M Jensen, Principal Investigator — University of Southern Denmark
Locations (1):
- University of Southern Denmark, Odense, Denmark

IPD SHARING:
Plan to Share IPD: Undecided